CLINICAL TRIAL: NCT04367610
Title: Effects of A Standardized Treatment Approach Comprising Plasma Exchange, Intravenous Immunoglobulin and Rituximab on Kidney Transplant Recipients With Acute or Chronic Antibody-Mediated Rejection
Brief Title: Effects of A Standardized Treatment Approach on Kidney Transplant Recipients With Antibody-Mediated Rejection
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Safak Mirioglu, Principal Investigator, Istanbul University
Other Study IDs: 2019/976
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Antibody-mediated Rejection; Kidney Transplant Rejection; Graft Loss
Keywords: antibody-mediated rejection; kidney transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Kidney transplant recipients with biopsy-proven acute or chronic antibody-mediated rejection who were treated using 6 sessions of therapeutic plasma exchange, 2 g/kg of intravenous immunoglobulin and 1-2 weekly doses of 375 mg/m2 rituximab.

SUMMARY:
Antibody-mediated rejection (ABMR) is one of the leading causes of graft loss in kidney transplant recipients (KTRs). Although it is a well characterized entity, there is limited data regarding effective treatment options for preserving graft functions. Moreover, results from different studies have been contradictory. Therefore, we conducted a study using our registry data to evaluate the effects of a standardized treatment approach consisting of therapeutic plasma exchange (regular plasmapheresis, double filtration plasmapheresis or immunoadsorption), intravenous immunoglobulin and rituximab on KTRs with acute or chronic ABMR.

ELIGIBILITY:
Inclusion Criteria:

* Being a kidney transplant recipient with biopsy-proven acute or chronic antibody-mediated rejection who were treated using 6 sessions of therapeutic plasma exchange, 2 g/kg of intravenous immunoglobulin and 1-2 weekly doses of 375 mg/m2 rituximab.

Exclusion Criteria:

* Not providing or withdrawing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients with biopsy-proven acute or chronic antibody-mediated rejection who were treated using 6 sessions of therapeutic plasma exchange, 2 g/kg of intravenous immunoglobulin and 1-2 weekly doses of 375 mg/m2 rituximab.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Graft Loss | 2-5 years
  Returning to dialysis due to graft failure or death with a functioning graft.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Yazici, MD, Study Chair — Department of Internal Medicine, Istanbul Faculty of Medicine; Safak Mirioglu, MD, Principal Investigator — Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Djamali A, Kaufman DB, Ellis TM, Zhong W, Matas A, Samaniego M. Diagnosis and management of antibody-mediated rejection: current status and novel approaches. Am J Transplant. 2014 Feb;14(2):255-71. doi: 10.1111/ajt.12589. Epub 2014 Jan 8. PMID 24401076